CLINICAL TRIAL: NCT04723290
Title: SARS-CoV-2 Seroconversion Study Among GHdC Staff Members
Brief Title: COVID-19 Seroconversion Study Among GHdC Staff Members - Summer 2020
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grand Hôpital de Charleroi (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SERO-SARS-CoV-2 GHdC
Record Dates: First submitted 2021-01-21; First posted 2021-01-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Serologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serological tests (Experimental): All staff at GHdC who want to know their level of antibodies against SARS CoV-2
  Interventions: Diagnostic Test: Serological tests for SARS Cov-2

INTERVENTIONS:
Diagnostic Test: Serological tests for SARS Cov-2 — Each participant will have a blood test on a dry tube of maximum 8 ml of whole blood

SUMMARY:
The management of the Grand Hôpital de Charleroi hospital authorized the performance of a serology for each member of the establishment's staff in order to better characterize the proportion of its employees who have already been in contact with the SARS CoV-2 virus for organizational and evaluation purposes symptoms.

DETAILED DESCRIPTION:
At the start of the SARS-CoV-2 pandemic, several workers had symptoms compatible with COVID-19 at a time when PCR (smear) testing was only allowed for hospitalized people. In addition, the PCR test has a fairly low sensitivity. In this context, serology can make it possible to determine whether the symptoms are indeed linked to exposure to SARS-CoV-2.

As a hospital, and in order to prepare for a possible second epidemic wave, it is also useful to know the proportion of staff members who have already been in contact with the virus for organizational purposes and symptom assessment.

.

ELIGIBILITY:
Inclusion Criteria:

* Be a member of the staff of the Grand Hôpital de Charleroi who wishes to participate in order to know their immunity related to SARS CoV-2 after the first wave of pandemic.

Exclusion Criteria:

* Not be part of the staff of the Grand Hôpital de Charleroi.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2817 (Actual)
Dates: Start 2020-06-20 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Serological tests to know the level of antibodies against SARS CoV-2 | up to 6 weeks
  The hospital has organized several schedules and appointments for each staff member depending on the ability to analyze laboratory samples and blood draws.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie de Visscher, MD, Principal Investigator — Grand Hôpital de Charleroi
Locations (1):
- Grand Hôpital de Charleroi, Charleroi, Hainaut, Belgium

IPD SHARING:
Plan to Share IPD: No
At this moment, there is no plan to share the results

REFERENCES:
- [Derived] de Visscher N, Holemans X, Gillain A, Kornreich A, Lagasse R, Piette P, Ventura M, Thys F. SARS-CoV-2 Seroprevalence among Healthcare Workers after the First and Second Pandemic Waves. Viruses. 2022 Jul 14;14(7):1535. doi: 10.3390/v14071535. PMID 35891515